CLINICAL TRIAL: NCT04934813
Title: Clinical Evaluation of Different Alveolar Ridge Preservation Techniques After Tooth Extraction: a Single- Center, Triple Blinded Randomized Clinical Trial.
Brief Title: Alveolar Ridge Preservation Techniques After Tooth Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Iosif El-Sioufi, Principal investigator, Iosif El-Sioufi, Master of Science in Periodontology, School of Dentistry, National and Kapodistrian University of Athens, National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Ethical committe No324
Record Dates: First submitted 2021-06-04; First posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-06

CONDITIONS: Alveolar Bone Loss
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Alveolar ridge preservation with particulated allograft covered with collagen sponge. (Experimental): Alveolar ridge preservation after tooth extraction. Freeze-dried bone allograft (FDBA) was applied in the socket immediatelly after tooth extraction and it was covered with collagen sponge (CS).
  Interventions: Other: Alveolar ridge preservation
- Alveolar ridge preservation with particulated allograft covered with autogenous soft tissue punch (Experimental): Alveolar ridge preservation after tooth extraction. Freeze-dried bone allograft (FDBA) was applied in the socket immediatelly after tooth extraction and it was covered with free gingival graft (FGG).
  Interventions: Other: Alveolar ridge preservation
- Alveolar ridge preservation with particulated xenograft covered with autogenous soft tissue punch (Experimental): Alveolar ridge preservation after tooth extraction. Demineralized bovine bone mineral xenograft (DBBM) was applied in the socket immediatelly after tooth extraction and it was covered with free gingival graft (FGG).
  Interventions: Other: Alveolar ridge preservation
- Alveolar ridge preservation without bone grafting covered with socket sealing mean (Experimental): Alveolar ridge preservation after tooth extraction. No bone graft was applied and the socket was covered with free gingival graft (FGG).
  Interventions: Other: Alveolar ridge preservation

INTERVENTIONS:
Other: Alveolar ridge preservation — application of different bone graft and sealing means after tooth extraction

SUMMARY:
The aim of the present randomized controlled trial (RCT) was to evaluate the efficacy of different alveolar ridge preservation (ARP) techniques on hard tissue dimensional alterations after tooth extraction, based on clinical measurements.

DETAILED DESCRIPTION:
Thrirty-six patients were randomly assigned in four treatment groups: A) freeze-dried bone allograft (FDBA) covered with collagen sponge (CS), B) FDBA covered with free gingival graft (FGG), C) demineralized bovine bone mineral xenograft (DBBM) covered with FGG and D) FGG without socket grafting. Clinical measurements were performed immediately after tooth extraction and 4 months later. The related outcomes pertained to both vertical and horizontal assessment of bone loss

ELIGIBILITY:
Inclusion Criteria:

* systematically healthy patients
* non-smokers
* no use of antibiotics for the last 3 months
* presence of a non-restorable single-rooted tooth in the maxilla.

Exclusion Criteria:

* Patients were excluded when a bony wall loss of more than 50% was verified for the socket after the extraction

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2019-12-20 (Actual); Study Completion 2020-06-25 (Actual)

PRIMARY OUTCOMES:
Vertical dimensional alterations of the alveolar ridge, after tooth extraction. | 4 months
  Assessment of the alteration of the alveolar ridge height after different alveolar ridge preservation techniques, based on clinical measurements. Clinical measurements were carried out immediately after tooth extraction and 4 months later. Distances in those clinical measurements were recorded in 0.1 mm increments, using a digital calliper (Logilink digital caliper WZ0031).
Horizontal dimensional alterations of the alveolar ridge, after tooth extraction. | 4 months
  Assessment of the alteration of the alveolar ridge width after different alveolar ridge preservation techniques, based on clinical measurements. Clinical measurements were carried out immediately after tooth extraction and 4 months later. Distances in those clinical measurements were recorded in 0.1 mm increments, using a digital calliper (Logilink digital caliper WZ0031).

CONTACTS AND LOCATIONS:
Locations (1):
- National and Kapodistrian University, Athens, Attica, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] El-Sioufi I, Oikonomou I, Koletsi D, Bobetsis YA, Madianos PN, Vassilopoulos S. Clinical evaluation of different alveolar ridge preservation techniques after tooth extraction: a randomized clinical trial. Clin Oral Investig. 2023 Aug;27(8):4471-4480. doi: 10.1007/s00784-023-05068-1. Epub 2023 May 25. PMID 37227497